CLINICAL TRIAL: NCT07217028
Title: Study Evaluating [18F]NOTA-ABY030 for Safety and Tolerability of Indeterminate Primary and/or Metastatic Disease in Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Eben Rosenthal, Barry and Amy Baker Professor and Department Chair, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: VICCHNP25055
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: SCC - Squamous Cell Carcinoma; Radiotracer; Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma
Keywords: unknown primary; cancer; hnscc; scc
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — Cetuximab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Dosimetry (3 Whole Body PET/CT Scans) (Experimental): Cohort A will include a minimum of six participants up to 12 participants. These participants will receive a 50 mg intravenous infusion of cetuximab, followed by a bolus injection of [18F]NOTA-ABY-030 at a dose of 5 (±1) mCi. To evaluate tracer distribution and radiation exposure, participants in this cohort will undergo three whole-body PET/CT scans at specific timepoints: 0-90 minutes, 120 minutes, and 240 minutes post-injection. Each scan will cover the region from the skull to mid-thigh, with a total imaging time of approximately 90 minutes. This cohort is essential for determining the absorbed dose, organ-specific uptake, identification of critical organs, and the effective dose of the radiopharmaceutical. The data collected from Cohort A will inform safety parameters and support dose optimization for future clinical studies involving [18F]NOTA-ABY-030.
  Interventions: Drug: Cetuximab (EGFR inhibitor); Drug: 18F-NOTA-ABY-030; Procedure: Positron Emission Tomography (PET)
- Cohort 2 - (1 Whole Body PET/CT Scan) (Experimental): Cohort 2 will include 54 participants. Each participant will receive a 50 mg intravenous infusion of cetuximab, followed by a bolus injection of [18F]NOTA-ABY-030 at a dose of 5 (±1) mCi. Imaging for this cohort will be conducted at a single timepoint, approximately 0-240 minutes (±15 minutes) post-injection, based on optimized timing derived from Cohort 1 data. The PET/CT scan for Cohort 2 will cover the region from skull to chest, with a total scan time of approximately 30 minutes. This cohort is designed to evaluate the diagnostic performance of [18F]NOTA-ABY-030 in identifying indeterminate metastatic and/or primary lesions in head and neck squamous cell carcinoma (HNSCC), with a focus on sensitivity, specificity, and feasibility of the imaging protocol in a broader patient population.
  Interventions: Drug: Cetuximab (EGFR inhibitor); Drug: 18F-NOTA-ABY-030; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Cetuximab (EGFR inhibitor) — Given IV
Drug: 18F-NOTA-ABY-030 — Given Bolus Injection
Procedure: Positron Emission Tomography (PET) — Undergo PET/CT

SUMMARY:
This Phase I, single-institution, open-label study will evaluate the safety, tolerability, and diagnostic performance of [18F]NOTA-ABY030 PET/CT in patients with head and neck squamous cell carcinoma (HNSCC) who present with indeterminate lesions on standard imaging. The investigational agent is a radiolabeled anti-EGFR affibody designed for rapid clearance and improved tumor-to-background contrast. All participants will receive a 50 mg cetuximab loading dose followed by a bolus of [18F]NOTA-ABY030, with PET/CT imaging performed at defined intervals to assess biodistribution and lesion uptake. The primary objective is to determine safety and tolerability; secondary objectives include radiation dosimetry and comparison of sensitivity and specificity to conventional imaging modalities (MRI, CT, and [18F]FDG-PET/CT). This approach aims to improve diagnostic accuracy, reduce unnecessary biopsies, and streamline treatment decisions for patients with HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subjects diagnosed with any T stage, any subsite within the head and neck. Subjects with recurrent disease or a new primary will be allowed.
3. Must have evidence of indeterminate metastatic and/or primary SCC based on clinical imaging or Primary SCC with suspicious Lymph Nodes standard image modalities prior to surgical removal
4. Have acceptable lab values, including the following clinical results (if values are considered clinically significant per investigator, participants must be asymptomatic):

   1. Hemoglobin ≥ 9gm/dL
   2. White blood cell count > 3000/mm3
   3. Platelet count ≥ 100,000/mm3
   4. Serum creatinine ≤ 1.5 times upper reference range
   5. Potassium
   6. Magnesium
   7. Phosphorus

Exclusion Criteria:

1. Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment.
2. Prior severe infusion reactions or hypersensitivity to other monoclonal antibody therapies.
3. Pregnant (based on Screening serum or urine pregnancy test administered before infusions), or breastfeeding.
4. Participants with known hypersensitivity to NOTA-ABY-030, cetuximab, murine, or any of the drug components used in this trial.
5. Subjects with history or evidence of interstitial pneumonitis or pulmonary fibrosis.
6. Severe renal disease or anuria.
7. Participants presenting with a baseline QTcF interval > than 480 milliseconds.
8. Those with an allergy to red meat, a history of tick bites, and alpha-gal syndrome will be given extra consideration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Assess number, grade and severity of adverse events to determine safety and tolerability of [18F]NOTA-ABY-030 in human subjects. | From infusion to 7 days post-infusion
  As determined by the number of adverse events (AEs) that are possibly or probably related to the study drug within 24 hours after infusion. Dose limiting toxicities will be defined as an AE grade >2 that is clinically significant and attributable to the study drug.

SECONDARY OUTCOMES:
Determination of the radiation dosimetry for [18F]NOTA-ABY-030 in human subjects. | From infusion to 7 days post-infusion
  The dosimetry for [18F]NOTA-ABY-030 will be determined to be the absorbed dose, organ specific uptake, critical organs, and effective dose for this first-in-human radiopharmaceutical.
Compare sensitivity and specificity of standard of care imaging modalities (MRI, CT, and/or [18F]FDG PET/CT) to [18F]NOTA-ABY-030-PET/CT for detection of indeterminate metastatic and/or primary lesion(s) in HNSCC | From infusion to 7 days post-infusion
  The specificity and sensitivity of [18F]NOTA-ABY-030 will be compared to the specificity and sensitivity of standard of care imaging obtained (MRI, CT, and/or [18F]FDG PET/CT) for identification of metastatic or primary lesion.

OTHER OUTCOMES:
Determine the sensitivity and specificity of [18F]NOTA-ABY-030 for the detection of indeterminate metastatic and/or primary lesion(s) in HNSCC. | From day of infusion to 36 months post-infusion
  The total number of HNSCC accurately detected by [18F]NOTA-ABY-030 compared to the number of positive disease during the 36 ± 6-month follow-up period (gold standard).

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not plan to share individual participant data from this phase 1 study due to its exploratory nature with a new drug. Sharing individual-level data at this stage could compromise participant confidentiality and may not yield meaningful insights given the preliminary scope of the study. Additionally, the data collected may not meet the robustness or generalizability standards required for broader dissemination. The investigators do not plan to share IPD with other researchers at this time.